CLINICAL TRIAL: NCT00477204
Title: Clinical Trial of Zocor and Vytorin in Adolescents With Type 1 Diabetes
Brief Title: Clinical Trial of Zocor (Simvastatin) and Vytorin (Ezetimibe/Simvastatin) in Adolescents With Type 1 Diabetes
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry); National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 06-1036; K23DK075360 (NIH)
Record Dates: First submitted 2007-05-21; First posted 2007-05-22 (Estimated); Results first posted 2013-06-21 (Estimated); Last update posted 2020-11-10 (Actual); Status verified 2020-10

CONDITIONS: Type 1 Diabetes Mellitus; Dyslipidemia
Keywords: Type 1 Diabetes Mellitus; dyslipidemia; adolescents
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Dyslipidemias | interventions — Simvastatin; Ezetimibe, Simvastatin Drug Combination

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Simvastatin (Active Comparator): Zocor(simvastatin)(20 mg)daily for 6 months along with Placebo (sugar pill)of active comparator (Vytorin [simvastatin] + Zetia [ezetimibe].
  Interventions: Drug: Simvastatin
- Ezetimibe/Simvastatin (Active Comparator): Vytorin(simvastatin [Zocor} + ezetimibe [Zetia])(20 mg)daily for 6 months along with placebo (sugar pill)of comparator (Vytorin [simvastatin]).
  Interventions: Drug: Ezetimibe/Simvastatin

INTERVENTIONS:
Drug: Simvastatin — simvastatin 20 mg daily
  Other Names: Zocor
  Arms: Simvastatin
Drug: Ezetimibe/Simvastatin — Ezetimibe (10mg)/Simvastatin (20mg)
  Other Names: Vytorin
  Arms: Ezetimibe/Simvastatin

SUMMARY:
The purpose of the study is to establish the safety of ezetimibe/simvastatin and simvastatin in adolescents with Type 1 Diabetes and to determine the amount of decrease in LDL-cholesterol.The study hypothesizes that simvastatin and ezetimibe/simvastatin will be safe in adolescents with Type 1 Diabetes and will lower LDL-cholesterol at 6 months.

DETAILED DESCRIPTION:
Cardiovascular disease is the leading cause of death in people with type 1 diabetes mellitus (T1DM) and since atherosclerosis begins in childhood, data to inform clinicians as to appropriate dyslipidemia treatment in this high-risk population are of great public health importance. In this trial of lipid-lowering medications (Zocor [simvastatin], a statin, compared to Vytorin [ezetimibe/simvastatin], a combination of a statin and Zetia, a medication that blocks cholesterol absorption) will be performed in patients ages 12-18 years with LDL ≥ 130 mg/dl, consistent with current ADA guidelines. The study hypothesizes that Zocor and Vytorin will be safe in adolescents with T1DM and will lower LDL-cholesterol at 6 months compared to baseline. In a two-arm design, Vytorin will lower LDL-c more than monotherapy with Zocor.

ELIGIBILITY:
Inclusion Criteria:

* 12-18 years of age with Type 1 Diabetes and seen at the Barbara Davis Center for Childhood Diabetes
* Positive diabetes auto-antibodies or provider diagnosed Type 1 Diabetes
* LDL > 130 mg/dl.

Exclusion Criteria:

* Familial hypercholesterolemia, Triglycerides (TG) > 400mg/dl
* Type 1 Diabetes of less than three-month duration
* HbA1c>9.5%
* Abnormal thyroid function
* Abnormal Creatine Kinase (CK) values (defined as > 10 times the upper limit of normal)
* Abnormal liver function tests (ALT/AST) (defined as >3 times the upper limit of normal)
* Pregnancy, and patients on oral contraceptives
* All resources are in English. Spanish speakers will not be available for the follow-up calls.

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 9 (Actual)
Dates: Start 2007-05; Primary Completion 2010-08 (Actual); Study Completion 2010-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David M Maahs, MD, Principal Investigator — University of Colorado, Denver; R. P Wadwa, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Barbara Davis Center for Childhood Diabetes, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Dates of recruitment: baseline 12/20/07-2/9/10; all participants completed 6-month trial by 8/3/10. All study participants seen at a medical clinic in an area designated for clinical research.
Pre-assignment Details: We identified 105 potential subjects. Of these, 42 patients proved to be ineligible, 26 declined invitation to a screening visit, 16 were not able to be scheduled, and 3 were interested but ineligible for the study. Therefore, 18 agreed to be in the study and 17 subjects attended a study screening visit of which 9 were enrolled in the study.
Groups:
- Ezetimibe/Simvastatin: ezetimibe/simvastatin : ezetimibe/simvastatin 10/20 mg daily placebo for each medication
- Simvastatin: simvastatin: simvastatin 20 mg daily
  placebo for each medication
Period: Overall Study
Arm/Group | Ezetimibe/Simvastatin | Simvastatin
Started | 4 | 5
Completed | 4 | 5
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Vytorin; Zocor: simvastatin, ezetimibe/simvastatin : simvastatin 20 mg daiy ezetimibe/simvastatin 10/20 mg daily placebo for each medication
- Total: Total of all reporting groups
Arm/Group | Vytorin | Zocor | Total
Number analyzed (Participants) | 4 | 5 | 9
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 4 | 5 | 9
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 13.7 (1.8) | 17.5 (2.3) | 15.8 (2.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 3 | 4
  Male | 3 | 2 | 5
Region of Enrollment [Number; unit: participants]
  United States | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: Change in LDL-c From Baseline to 6 Months in Subjects With Type 1 Diabetes Taking Vytorin or Zocor.
Description: Change in LDL-c between Zocor and Vytorin treatment in subjects with Type 1 Diabetes measured at baseline to the 6-month study visit.
Time Frame: Baseline to 6 months
Population: Recruitment for this study failed to meet target. Due to the small sample size the analyses of these data were primarily descriptive.
Measure: Mean (Standard Deviation); unit: mg/dl
Groups:
- Vytorin (Ezetimibe/Simvastatin): ezetimibe/simvastatin : ezetimibe/simvastatin 10/20 mg daily placebo for each medication
- Zocor (Simvastatin): simvastatin: simvastatin 20 mg daily
  placebo for each medication
Arm/Group | Vytorin (Ezetimibe/Simvastatin) | Zocor (Simvastatin)
Number analyzed (Participants) | 4 | 5
mg/dl | -67 (47) | -6 (25)

ADVERSE EVENTS:
Time Frame: All Serious Adverse Events (SAEs) will be reported to the Clinical Translational Research Center (CTRC), Data Safety Monitoring Board (DSMB), Research Subject Advocate (RSA) and the Colorado Multiple Institutional Review Board (COMIRB) within 5 days
Description: SAEs will also be reported to the FDA since this protocol is under an Investigational New Drug (IND). Adverse Events (AEs) will be batched and reported to the DSMB as part of the periodic reports and to COMIRB at the time of continuing review.
Groups:
- Vytorin (Simvastatin + Ezetimibe): Vytorin [simvastatin + ezetimibe]20 mg taken daily for 6 months to compare in a 2- arm design to Zocor [simvastatin] .
- Zocor [Simvastatin]: Zocor [simvastatin] 20 mg taken daily for 6 months to compare in a 2- arm design to Vytorin [simvastatin + ezetimibe].
Arm/Group | Vytorin (Simvastatin + Ezetimibe) | Zocor [Simvastatin]
Serious Adverse Events (participants affected / at risk) | 0/4 | 0/5
Other Adverse Events (participants affected / at risk) | 0/4 | 0/5

LIMITATIONS AND CAVEATS:
Recruitment for this study failed to meet target and therefore it is difficult to make conclusions on the data obtained in these 9 subjects. No secondary outcomes were measured as recruitment was insufficient and study was stopped after only 9 subjects completed trial.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The only disclosure restriction on the PI is that the sponsor can review results communications prior to public release and can embargo communications regarding trial results for a period that is less than or equal to 30 days from the time submitted to the sponsor for review.